CLINICAL TRIAL: NCT01724970
Title: A Randomized Comparative Study on Proseal LMATM and Supreme LMATM for Bariatric Surgery.
Brief Title: Laryngeal Masks for Bariatric Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2276P
Record Dates: First submitted 2012-09-14; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Morbid Obesity
Keywords: anesthesia; postanesthetic recovery; ventilation; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLMA (Experimental): ProSeal
  Interventions: Device: ProSeal
- SLMA (Experimental): Supreme LMA
  Interventions: Device: Supreme LMA

INTERVENTIONS:
Device: ProSeal — Patients will be ventilated with PLMA
  Arms: PLMA
Device: Supreme LMA — Patients will be ventilated with SLMA
  Arms: SLMA

SUMMARY:
Obese people pose specific problems as far as the management of airway during surgery. The study aims to compare efficacy and safety of two LMA devices.

DETAILED DESCRIPTION:
The study will investigate two types of LMA devices endowed of different constructive features. The two devices share common features as far as providing access to the stomach and reducing morbidity of the upper airway. The two device differ in regard to ease of insertion and sealing of the airway and these features are particularly important in the obese patient.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III
* candidates to bariatric surgery

Exclusion Criteria:

* uncontrolled psychiatric symptomatology
* known or presumed pregnancy
* history of surgery on the airway or esophagus
* gastroesophageal reflux

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | intraoperatively, up to 3 hours

SECONDARY OUTCOMES:
total anesthetic and analgesic drug dosages | intraoperatively and postoperatively, up to 24 hours from end of surgery
pulse oximetry saturation | intraoperatively and postoperatively, up to 24 hours from end of surgery
time to post-anesthetic discharge scoring system (PADSS) > 8 | in PACU up 72 hours
EKG monitoring | postoperatively up to 72 hours
satisfaction of the surgeon (ad hoc questionnaire) | day 1
satisfaction of the patient (Iowa Satisfaction with Anesthesia Scale) | day 1
gastric distension | intraoperatively up to 3 hours
levels of pain and nausea (Visual Analogue Scale) | postoperatively up to 24 hours
metilen's blue | before end of surgery up to 3 hours
total dosage of analgesic and antihemetic drugs | intra and postoperatively up to 24 hours

OTHER OUTCOMES:
insertion time | up to 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michele Carron, MD, Principal Investigator — University of Padova
Locations (1):
- University of Padua, Padua, PD, Italy